CLINICAL TRIAL: NCT03680768
Title: Development of a New Biological Age Technology Applicable in Public Health Promotion Interventions.
Brief Title: Biological Age in Health Promotion - Novel Health Technology
Acronym: BATE
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Jørn Wulff Helge, Ph.D., Proffesor Jørn Wulff Helge, University of Copenhagen
Other Study IDs: Biological Age Technology
Record Dates: First submitted 2018-09-17; First posted 2018-09-21 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Aging; Healthy
Keywords: Health; Risk of disease; Prediction; Lifestyle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample will be drawn from a vein in the elbow
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Health Assessment — The protocol includes measurements of body composition, strength test, functional and fitness test as well as biochemical measurements from blood samples and AGEreader

SUMMARY:
The purpose of this cross-sectional study is to collect relevant molecular markers of aging and measures of physiological function. Together these biomarkers are used to develope a new Biological Age model, useful in health promotion interventions in the public health sector .

DETAILED DESCRIPTION:
Study design: 100 participants representing the healthy danish working adult population. This study seek to include both men and women equally distributed in the range of 18-65 of age.

Data collection: After recruitment, participants need to attend once to the laboratory, overnight fasted and without having exercised for the previous 24 hours.

All analyse are done in investigators lab (Xlab) at the department of Biomedical Sciences, Copenhagen University. When analyzes are done, the results are used in algorithm developement in cooperation with Technical university Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Males and females interested in their personal health status
* Healthy males and females

Exclusion Criteria:

* Pregnancy
* Previous or current cardiovascular disease
* Use of medication that affects our measurements such as betablockers,statins or medication that affects the metabolism.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sample size representing the general healthy danish population
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Biological Age | Day 1
  A composite score of ones biological state (in years)

SECONDARY OUTCOMES:
Fitness Level | Day 0
  VO2max - maximal oxygen consumption (ml/min/kg)
Strength | Day 0
  Hand grip, isometric quadriceps and biceps strength (Nm)
Sit to Stand test | Day 0
  Rise and sit from a chair as many times as possible during 1 minute (number og rises)
Central obesity | Day 0
  Waist to hip ratio is measured by dividing waist circumference with hip circumference in cm.
Weight | Day 0
  measured in kilograms
Height | Day 0
  measured in cm
Body composition | Day 0
  BMI (kg/m2) is calculated
Muscle mass | Day 0
  muscle mass(g) is assessed by dual energy x-ray absorptiometry (DXA) and bioimpedance
Fat mass | Day 0
  fat mass(g) is assessed by DXA and bioimpedance
Fat percentage | Day 0
  Fat%, is assessed by DXA and bioimpedance
Lipid profile | Day 0
  HighDensityLipoprotein (mmol/L), LowDensityLipoprofile (mmol/L), TriGlycerides (mmol/L), FreeFattyAcids (mmol/L) and Glycerol (mmol/L) is measured in a blood sample.
Hormones | Day 0
  Sex hormones: testosteron and estradiol (nmol/L) and InsulinGrowthFactor-1 (nmol/L) and Insulin (µU/ml) ais analysed from blood samples
Inflammatory profile | Day 0
  C-reactive protein mg/L, soluble urokinase plasminogen activating receptor ng/ml, InterLeukin 6,8 and 10 (pg/mL), tumor necrosis factor (pg/mL), Leptin and Adiponectin (ng/ml) is analysed from blood samples
Levels of glycated protein and lipids as a result of exposure of excess sugars | Day 0
  advanced glycation endproducts (AGE) measured in the skin
Color passport photography | Day 0
  Profile picture taken to assess perceived age
Respirometry | Day 0
  forced vital capacity and forced expiratory volume at one second(L)
Blood Pressure | Day 0
  Systolic and Diastolic blood pressure (mmHg)
Blood glucose | Day 0
  HbA1c and fasting glucose (mmol/L) measured from blood sample
Blood profile | Day 0
  Haematocrit and Haemoglobin (mmol/L) measured in a blood sample
Aging biomarker | Day 0
  Chemokines Eotaxin (CCL11) analysed from blood samples
Youth biomarker | Day 0
  Growth Differential Factor (GDF-11) analysed from blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Jørn W Helge, Prof, Principal Investigator — Biomedicinsk Institut
Locations (1):
- University of Copenhagen, Department of Biomedical Sciences, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Husted KLS, Brink-Kjaer A, Fogelstrom M, Hulst P, Bleibach A, Henneberg KA, Sorensen HBD, Dela F, Jacobsen JCB, Helge JW. A Model for Estimating Biological Age From Physiological Biomarkers of Healthy Aging: Cross-sectional Study. JMIR Aging. 2022 May 10;5(2):e35696. doi: 10.2196/35696. PMID 35536617
- [Derived] Husted KLS, Fogelstrom M, Hulst P, Brink-Kjaer A, Henneberg KA, Sorensen HBD, Dela F, Helge JW. A Biological Age Model Designed for Health Promotion Interventions: Protocol for an Interdisciplinary Study for Model Development. JMIR Res Protoc. 2020 Oct 26;9(10):e19209. doi: 10.2196/19209. PMID 33104001